CLINICAL TRIAL: NCT01066455
Title: PITT1109: Cardiac Outcome Measures in Children With Muscular Dystrophy
Brief Title: Cardiac Outcome Measures in Children With Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: PITT1109
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Limb Girdle Muscular Dystrophy
Keywords: Cardiac; Muscular Dystrophy; Prospective; Pediatric; Echocardiogram
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies, Limb-Girdle; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Prospective collection of blood sample for BNP measurements.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the research study is to evaluate different cardiac measures that are obtained by echocardiographic tests in patients with muscular dystrophy.

DETAILED DESCRIPTION:
The research study will include 50 participants aged 8 to 18 years old (before 18th birthday) with Duchenne, Becker, or autosomal recessive limb-girdle (specifically: LGMD 2C-2F and 2I) muscular dystrophies.

Participants will be seen in one of five Cooperative International Neuromuscular Research Group (CINRG) centers located in the United States.

All study assessments will be completed in the same day and include reviewing past medical and surgical history, collecting vital signs, collecting cardiac measures through echocardiographic tests.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 8 and 18 years old
* Confirmed diagnosis of muscular dystrophy (DMD, BMD, or LGMD 2C-2F and 2I)

Exclusion Criteria:

* Investigator assessment of inability to comply with protocol
* History of a congenital cardiac defect or other cardiac disease unrelated to muscular dystrophy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 8 to 18 years old Confirmed diagnosis of Duchenne, Becker, or autosomal recessive limb-girdle muscular dystrophy (LGMD: 2C-2F and 2I)
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California Davis, Sacramento, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington University St. Louis, St Louis, Missouri
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas